CLINICAL TRIAL: NCT02002858
Title: Integrated Smoking Cessation Treatment for Emotional Dysregulation
Brief Title: Smoking Cessation for Depression and Anxiety Treatment
Acronym: SDAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA03474101; R34DA034741 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-06 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Smoking; Anxiety Disorders; Depression Disorders
Keywords: smoking; cessation; anxiety; anxious; depression; depressed; smoker; stress
MeSH Terms: conditions — Smoking; Anxiety Disorders; Depression; Consciousness Disorders | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depression and Anxiety Smoking Cessation Treatment (Experimental): Cognitive-behavioral treatment program that blends smoking cessation, anxiety, and depression management/reduction treatment strategies
  Interventions: Drug: Nicotine Patch; Behavioral: Depression and Anxiety Smoking Cessation Treatment
- Educational-Support Psychotherapy (Active Comparator): Educational-based psychotherapy and standard smoking cessation treatment program
  Interventions: Drug: Nicotine Patch; Behavioral: Educational-Support Psychotherapy

INTERVENTIONS:
Drug: Nicotine Patch
Behavioral: Depression and Anxiety Smoking Cessation Treatment — Cognitive-behavioral treatment program that blends smoking cessation, anxiety, and depression management/reduction treatment strategies
  Other Names: SDAT
  Arms: Depression and Anxiety Smoking Cessation Treatment
Behavioral: Educational-Support Psychotherapy — Educational-based psychotherapy and standard smoking cessation treatment program
  Arms: Educational-Support Psychotherapy

SUMMARY:
The primary aim of this research study is to enhance smoking cessation outcome among smokers with elevated anxiety and depression. We are comparing two group treatment approaches: (1) An educational-supportive psychotherapy and standard smoking cessation treatment, and (2) An integrated smoking cessation, and anxiety and depression management treatment program (SDAT). Both treatments also utilize nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years old
* Capable of providing informed consent
* Willing to attend all study visits and comply with the protocol
* Daily smoker for at least one year
* Currently smoke an average of at least 6 cigarettes per day
* Report a motivation to quit smoking in the next 6 weeks of at least 5 on a 10-point scale
* Elevated anxiety or depression

Exclusion Criteria:

* Use of other tobacco products
* Current or past psychotic disorders of any type, or comorbid psychiatric conditions that are relative or absolute contraindications to the use of any treatment option in the study protocol
* Currently suicidal or high suicide risk
* Current use of any pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt
* Concurrent psychotherapy initiated within three months of baseline, or ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety or depression
* Current or intended participation in a concurrent substance abuse treatment
* Current non-nicotine substance dependence
* Insufficient command of English to participate in assessment or treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Smoking Status using the Timeline Follow-Back Assessment | Change from baseline at 2, 4, 8, 10, 16, and 24 weeks post quit day.
  Participants will report the number of cigarettes they consumed everyday since their last visit. The number of cigarettes reported will be used to determine smoking status (e.g., 0 cigarettes reported is abstinent and any cigarettes reported is currently smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Laboratory and Substance Use Treatment Clinic, Houston, Texas, United States